CLINICAL TRIAL: NCT02297282
Title: A Pragmatic Randomized Trial to Investigate the Effectiveness of BehaviouRal ActiVation Group Therapy in Reducing dEpressive Symptoms and Improving Quality of Life in Patient With Depression: BRAVE Study.
Brief Title: A Study to Assess the Effectiveness of Behavioural Activation Group Therapy in Individuals With Depression
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Zainab Samaan (Zena), Associate Professor and Psychiatrist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVE_Main Study
Record Dates: First submitted 2014-09-05; First posted 2014-11-21 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Depression
Keywords: Depression; Behavioural Activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioural Activation (Experimental): Originally a component of Cognitive Therapy, behavioural activation is the use of strategies such as activity scheduling, master/pleasure ratings, and graded task assignments to change one's perception of specific situations. Behavioural Activation involves the use of activities to improve life situations or depressed mood.
  Interventions: Behavioral: Behavioural Activation (BA)
- Wait List (Control Group) (No Intervention): The Control group (waitlist) will receive treatment as usual while they are waiting to start the BA intervention at the end of the Intervention Group Therapy time (28 sessions over an 18 week period). In addition to usual care, the control group will be assessed by clinical staff that offers treatment as usual for mood symptoms and quality of life measures during the waiting time.

INTERVENTIONS:
Behavioral: Behavioural Activation (BA) — Behavioural activation is a therapy, which has been shown to be quite effective in the treatment of depression. Originally a component of cognitive therapy, behavioural activation is the use of strategies such as activity scheduling, master/pleasure ratings, and graded task assignments to change one's perception of specific situations. It involves the use of activities to improve life situations or depressed mood.
  Arms: Behavioural Activation

SUMMARY:
Depression affects 15% of Canadians resulting in serious impact on health, ability to function including social, family and work related activities. Despite the several treatment options available for managing depression including medications, many patients do not respond to treatment and experience troublesome side effects. Psychotherapies are important in the treatment of depression and several options are currently being offered at the Mood Disorders Program (MDP), St. Joseph's Healthcare Hamilton. However a simple and reportedly effective therapy called Behavioural Activation (BA) is not currently available and existing evidence supporting its' effectiveness is limited to individual therapy of community based patients who are unlike the patients seen at the MDP who may have a more severe illness. The investigators are therefore planning to study the effectiveness of BA in patients with depression as an add on therapy to existing usual care compared to wait-list added to usual care. The study outcome is reduction in depressive symptoms and improvement in quality of life. The duration of therapy is 18 weeks and all adults with depression are eligible to participate.

DETAILED DESCRIPTION:
This study is a pragmatic randomized controlled trial to test the effectiveness of behavioural activation in depression. The pragmatic randomized controlled trial study design is a parallel 1:1 allocation comparing behavioural activation plus treatment as usual to waitlist control group plus treatment as usual. For this study the investigators will adopt the following principals simulating naturalistic real life clinical setting to test the study question based on the pragmatic design:

1. No restrictive inclusion criteria will be used. Adults with major depressive disorder will be asked to participate in this study
2. Clinicians will deliver the BA program to participants randomized to receive the intervention
3. The intervention will be an add-on to treatment as usual
4. The comparison group will receive treatment as usual that may include medications, CBT and other therapies as required and decided by their clinical care
5. The primary outcome is clinically relevant (improvement in depressive symptoms and quality of life)
6. Both the intervention and control groups will be assessed as intention to treat analysis with no measures to improve adherence to the study intervention or the comparator.

Patients with a diagnosis of depressive disorders attending the mood disorders clinic, referred for assessment of depression at the clinic or referred from community or other hospital services to the mood disorders clinic will be approached for participation in the study. In addition family practices in the community will be informed of the study and asked to refer directly to the trial. Following initial screening for eligibility, potential participants will be asked to provide written informed consent prior to any study related procedures.

The investigators will employ a parallel group design to evaluate the effects of behavioural activation intervention to improve depression related outcomes. Eligible and consenting patients will be randomly allocated to the intervention or control arms using a 1:1 allocation ratio. Allocations will be generated using the computerized system. The randomization will use a block randomization system of block sizes of 2, 4 and 6. The assignment of participants to the intervention or control arms will be done after the screening visit and enrolment of at least 20 participants to ensure balanced groups. The allocation will be done by a research personnel who is not a clinician and will not know the participant clinical status to maintain allocation concealment.

This trial is an open label trial as blinding is not possible for participants (behavioural activation intervention) or the clinician administering the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder
* Must be able to provide written informed consent
* Must be able to attend program sessions

Exclusion Criteria:

* Inability to understand written and spoken English
* Primary diagnosis other than Major Depressive Disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2014-10; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Assess the effectiveness of a structured, therapist administered, face to face program of Behavioural Activation (BA) added to treatment as usual on depressive symptoms. | end of the study period (18 weeks)
  The Beck Depression Inventory (BDI-II) is administered to measure the effectiveness of BA on depressive symptoms.

SECONDARY OUTCOMES:
Test the effects of Behavioural Activation on changes in physical health parameters. | at end of the study period (18 weeks)
  Quality of life
Economic evaluation of the behavioural activation program in the study population. | at the study end point (18 weeks).
  Economic evaluation of the BA program will be assessed using the EuroQol 5-Dimension (EQ-5D-5L), a commonly used standardized generic measure of health status and quality of life in a variety of clinical conditions.

OTHER OUTCOMES:
A change in the mean weekly number of steps taken by participants. | up to 18 weeks
  Study participants within the BA arm will be provided with "Fitbit" activity tracking monitors for use during the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Samaan, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided